CLINICAL TRIAL: NCT05351866
Title: Feasibility and Acceptability of a Digital Therapeutic for Adolescent Depressive Symptoms in Hematology/Oncology and Weight Management
Brief Title: Digital Therapeutic for Adolescent Depressive Symptoms in Hematology, Oncology, and Weight Management
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low Enrollment
Sponsor: Limbix Health, Inc. (Industry)
Collaborators: Children's Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LMX-004
Record Dates: First submitted 2022-04-18; First posted 2022-04-28 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Depression; Depressive Disorder; Depressive Symptoms; Depressive Episode; Adolescent Behavior; Adolescent - Emotional Problem; Hematologic Diseases; Oncology; Weight, Body
Keywords: Depression; Mental Health; Adolescent mental health
MeSH Terms: conditions — Depression; Depressive Disorder; Adolescent Behavior; Hematologic Diseases; Neoplasms; Body Weight; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- SparkRx (Experimental): 5-week CBT-based mobile intervention for adolescents with depressive symptoms
  Interventions: Device: CBT-based mobile intervention for depression
- Educational Control (Active Comparator): 5-week mobile control with education about depression
  Interventions: Device: Mobile control with education about depression

INTERVENTIONS:
Device: CBT-based mobile intervention for depression — SparkRx is a 5-week program divided into levels intended to be completed weekly. SparkRx is a behavioral activation program. Participants are instructed to complete a weekly Patient Health Questionnaire (PHQ)-8 assessment and participant symptom check (PSC) in the mobile app. Tasks in the mobile app progress in a linear fashion (i.e., each task must be completed to progress to the next task).
  Other Names: SparkRx
  Arms: SparkRx
Device: Mobile control with education about depression — The control mobile application will consist of 5 weeks of educational content about depression. Participants will be instructed to complete a weekly Patient Health Questionnaire (PHQ)-8 assessment and PSC in the mobile app.
  Other Names: Educational Control
  Arms: Educational Control

SUMMARY:
The primary aims of the proposed research are to assess the feasibility, acceptability, and preliminary evidence of efficacy of a self-guided, cognitive behavioral therapy (CBT)-based mobile app intervention (SparkRx) for the treatment of adolescents presenting with symptoms of depression in specialty medical care settings (e.g.Hematology/Oncology, Weight Management, etc.) at Children's Health System of Texas (CHST).

DETAILED DESCRIPTION:
The primary aims of the proposed research are to assess the feasibility, acceptability, and preliminary evidence of efficacy of a self-guided, cognitive behavioral therapy (CBT)-based mobile app intervention (SparkRx) for the treatment of adolescents presenting with symptoms of depression in specialty medical care settings (e.g.Hematology/Oncology, Weight Management, etc.) at Children's Health System of Texas (CHST).

These aims will be accomplished by evaluating:

* Feasibility of recruiting and enrolling adolescents with mild to severe symptoms of depression from specialty care medical programs at CHST.
* Retention, program adherence, completion, and withdrawal rates.
* Perceived utility, usability, and enjoyment of the program by adolescents
* Clinically significant changes between pre- to -post treatment and persistence of such gains at 1 month follow up.
* Preliminary evidence of efficacy defined as a statistically significant difference in the eight-item Patient Health Questionnaire (PHQ-8) scores (p < 0.05) between Spark and an educational control at post-treatment.
* Safety of the intervention, including rates of reported adverse events and adverse device effects

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 13 and 22
* Moderate- severe self-reported symptoms of depression at baseline (PHQ-8 >= 5)
* Have a comorbid medical condition and under the care of a healthcare provider at CHST
* English fluency and literacy of adolescent; English or Spanish fluency and literacy of consenting legal guardian if under 18
* Access to a compatible smartphone (or other device) and operating system (i.e., capable of installing the app from the Google Play or Apple App Store; list will be provided to participants) and regular internet access
* Willing to provide informed consent/assent and have legal guardian willing to provide informed consent (if required)

Exclusion Criteria:

* Concurrent psychotherapy: Have met with a psychologist for intervention (not assessment) for 30 minutes or more, more than once in the 3 weeks prior to enrollment as determined by the study team
* Change in psychotropic medication (initiation or change in dose) within the past 30 days prior to enrollment
* Suicide attempt within the past year as determined at eligibility screening
* Active suicidal ideation with intent as determined at eligibility screening
* Previously participated in user testing or clinical testing of the Spark app
* Participating in any other psychiatric or psychological treatment based clinical research at the time of enrollment and up to two months prior to enrollment or planning to participate in any other psychiatric or psychological treatment based clinical research during the study intervention period (5 weeks)
* Any condition, comorbidity, or event that, in the opinion of the investigator, will prevent the participant from adhering to the protocol or benefiting from the treatment (e.g., unable to provide informed assent or consent) or will prevent investigators from being able to ensure safety (e.g., will be leaving the country during study time period)

Ages: 13 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Feasibility of intervention: Eligibility | Screening
  Percent of potential participants eligible to participate
Feasibility of intervention: Participant willingness | Screening
  Percent of eligible participants willing to participate
Feasibility of intervention: Completion adherence | 5 weeks
  Adherence to program determined by percent of enrolled participants completing all modules within 5 weeks and by post-treatment
Feasibility of intervention: Module adherence | 5 weeks
  Adherence to program determined by average number of modules completed
Feasibility of intervention: Time adherence | 5 weeks
  Adherence to program determined by engagement with program (time spent in app)

SECONDARY OUTCOMES:
Change in depressive symptoms | 5 weeks
  Measured by the Patient Health Questionnaire (PHQ-8). Score range of 0 to 24 with higher scores indicating worse outcome.
  * Clinically significant improvement: reduction in assessment score >= 5
  * Treatment response: 50% reduction in symptoms from pre to post-intervention
  * Remission is defined as a score < 5
Adverse events | 11 weeks
  Rates of adverse events and adverse advice effects
Usability | 5 weeks
  Usability measured with the System Usability Scale (SUS), which consists of 10 items, each with five response options for respondents; from Strongly agree to Strongly disagree. Scores range from 0-100, with higher scores meaning more usable.
Engagement | 5 weeks
  Engagement measured with the User Engagement Scale - Short Form (UES-SF), which measures self-reported user engagement. The form has 12 items and uses a 5 point Likert scale. Scores range from 1-5, with higher scores indicating more engaging material.

OTHER OUTCOMES:
Treatment-related change in depressive symptoms | Change over 5 weeks
  Difference in the change in PHQ-8 scores between the SparkRx and control arms. Score range of 0 to 24 with higher scores indicating worse outcome.
Treatment-related change in anxiety | Change over 5 weeks
  Measured by the Generalized Anxiety Disorder scale (GAD-7).The GAD-7 is a brief 7-item assessment for generalized anxiety disorder with satisfactory sensitivity and specificity. Score range of 0 to 21 with a higher score indicating worse outcome.
Treatment-related change in global functioning | Change over 5 weeks
  Measured using the Short Form-36 (SF-36), a set of generic, coherent, self-reported, and easily administered quality-of-life measures used to routinely monitor and assess the care outcomes of participants. 8 subscales with scores ranging from 0-100, higher being a more favorable health state.
  Physical functioning Role limitations due to physical health Role limitations due to emotional problems Energy/fatigue Emotional well-being Social functioning Pain General health
Caregiver proxy treatment-related change in depressive symptoms | Change over 5 weeks
  Measured using caregiver proxy measures of the PHQ-8. Score range of 0 to 24 with higher scores indicating worse outcome.
Caregiver proxy treatment-related change in global functioning | Change over 5 weeks
  Measured using caregiver proxy measures of the SF-36. 8 subscales with scores ranging from 0-100, higher being a more favorable health state.
Treatment-related change in hope | Change over 5 weeks
  Measured using the Hope Scale, a 12-item self-report measure, which assesses dispositional hope in adults. Each item rated from 1-8 (definitely false - definitely true). Scores range from 8-64, with higher being more hopeful.
  Subscales: agency and pathway.
Healthcare utilization | Change over 5 weeks
  Descriptive understanding of healthcare utilization. Measured by the Healthcare Utilization Questionnaire. A two-item questionnaire that assesses participants' use of healthcare resources.
Caregiver burden | Change over 5 weeks
  Descriptive understanding of caregiver burden, measured by the work absenteeism questionnaire, containing questions about caregiving responsibilities and related impacts on employment. Higher scores indicate more hours missed per week of work.
Treatment-related change in physical symptom severity | Change over 5 weeks
  Measured by the Functional Disability Inventory a fifteen-item questionnaire that measures functional disability and evaluates the impact of illness on the respondents' physical and psychosocial functioning in everyday social roles. Each question is rated on a 5-point scale from 0(No Trouble) to 4 (Impossible). Score range is 0 to 60 with higher scores indicating a worse outcome.
Treatment-related perceptions of experience with SparkRx | 5 weeks
  Measured by the User Experience (UXR) questionnaire. Includes questions from the Usability Metric for User Experience (UMUX)-Lite; a two-item questionnaire that assesses the usability of the mobile application. Questions have seven response options from Strongly agree to Strongly disagree. Includes questions from the Happiness Tracking Surveys (HaTs); an open-ended questionnaire that assesses respondents' experiences with the product and provides options for feedback.
Treatment expectations | 5 weeks
  Identifying the relationship between treatment expectations and treatment outcomes. Expectations measured with the Stanford Expectations of Treatment Scale (SETS), an instrument for measuring positive and negative treatment expectancies. There are two subscales, the positive and negative expectancy. Scores range from 1-7, with higher scores indicating greater positive and negative expectancy.
  Outcomes measured with the PHQ-8. Score range of 0 to 24 with higher scores indicating worse outcome.
Treatment expectations: Credibility/Expectancy | 5 weeks
  Identifying the relationship between treatment expectations and treatment outcomes. Expectations measured with the Credibility/Expectancy Questionnaire (CEQ), a questionnaire for measuring cognitively-based credibility and relatively more affectively-based expectancy of therapy outcomes. Scores range from 6-60, with higher scores indicating a greater expectation of treatment success.
  Outcomes measured with the PHQ-8. Score range of 0 to 24 with higher scores indicating worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Germann, PhD., Principal Investigator — Children's Health System of Texas
Locations (1):
- Children's Hospital Texas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No